CLINICAL TRIAL: NCT03696849
Title: Patient Satisfaction and Clinical Assessment of Surface Roughness and Wear of Enamel Antagonists for Polished Versus Glazed Posterior Lithium Disilicate Glass Ceramic Crowns
Brief Title: Clinical Assessement of Glazed Versus Polished Lithium Disilicate Crowns in Surface Roughness and Enamel Antagonists Wear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mervat Mourad Rouchdy Farid, assisstant lecturer, fixed prosthodontics department, faculty of oral and dental medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-09-34
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glazed emax Press (Active Comparator)
  Interventions: Other: polished emax Press
- Polished emax Press (Experimental)
  Interventions: Other: polished emax Press

INTERVENTIONS:
Other: polished emax Press — lithium disilicate glass ceramic crowns subjected to polishing only
  Other Names: emaxPressable ceramics

SUMMARY:
It is believed that final glazing yields the most acceptable ceramic surfaces in terms of smoothness. However, since reglazing must be performed in a dental laboratory with the use of a thermal furnace, it requires multiple office visits. Repeated firings have a destructive effect on ceramic surfaces and can cause deformation. Conversely, polishing is easy and simple and can be accomplished in a single session.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18-50 years old who are able to read and sign the informed consent document.
* Physically and psychologically able to tolerate conventional restorative procedures.
* Have no active periodontal or pulpal diseases, have teeth with good restorations.
* Patients have no temporomandibular disorders.
* Each participant needed a crown on either a first or second premolar or first or second molar in any arch.
* Teeth selected shoud include:

restorability with a crown:root ratio of at least 1:1. presence of an opposing natural tooth which was non-restored or minimally restored.

the presence of two non-restored or minimally restored teeth opposing each other on the same quadrants as the crowned tooth and the opposing to serve as enamel controls. Minimally restored was defined as teeth which have no restoration greater than a Class II amalgam restoration.

- Willing to return for follow-up examinations and evaluation.

Exclusion criteria

* Patients in the growth stage with partially erupted teeth.
* Patients with poor oral hygiene and motivation.
* Pregnant women.
* Psychiatric problems or unrealistic expectations.
* Lack of opposite occluding dentition in the area intended for restoration.
* Patients with temporomandibular disorders.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Antagonists enamel wear using profilometer | 1 year
  wear of enamel antagonists opposing to emaxPress crowns that will be measured in um

SECONDARY OUTCOMES:
Restoration surface Roughness using profilometer | 1 year
  restoration roughness after different finishing methods that will me measured in um
Patient satisfaction | 1 year
  Questionnaire